CLINICAL TRIAL: NCT03845803
Title: "Sit - Stand - Be Fit" - Influence of Sit/Stand Workstations on Sedentary Behaviour and the Prevalence and Intensity of Musculoskeletal Diseases in Office Workers of an Austrian Bank Headquarter
Brief Title: Reducing Sedentary Behaviour in Office Workers
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences for Health Professions Upper Austria (Other)
Responsible Party: Sponsor
Other Study IDs: A-2019-001
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Sedentary Lifestyle
Keywords: Sit/stand workstation; Office workers; Sedentary behaviour; Sitting time; Musculoskeletal disorder
MeSH Terms: conditions — Sedentary Behavior; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Reducing sedentary behaviour — Implementing sit/stand workstations at work

SUMMARY:
This is a one year observational field study investigating changes in sedentary behaviour and the prevalence of musculoskeletal disorders of office workers induced by sit/stand workstations. All employees of an Austrian bank headquarter (approx. 1200 people) will be newly equipped with electric sit/stand workstations by their company in February and March 2019. The main outcomes will be occupational sitting and standing time as well as the occurence and intensity of neck and back pain.

DETAILED DESCRIPTION:
Background Currently, 18.5 percent of all European Union citizens sit more than 7.5 hours per day. It is estimated that approximately one third of white-collar workers spend more than 7.5 hours per day seated. Moreover, it is assumed that working adults sit for up to two thirds of their working time on average, with some office-based occupations (e.g. call center employees) requiring workers to sit for more than 80% of their working day. Although the decline in physical activity helped to reduce physical overload and the accompanying risks, ongoing activity pattern changes are relevant factors in the development of health-related problems. Sedentary and sitting time are both risk factors for several diseases, such as obesity, depression and all-cause mortality. Interestingly, risks of prolonged sitting are independent of physical activity levels.

A possible way to reduce occupational sitting time are sit/stand workstations. Sit-to-stand workstations provide an incentive for people to work in either a sitting or standing posture and facilitate regular sit-to-stand transitions. Despite the global increase in incidence rates, the majority of office workers in Austria are still not provided with this kind of workstation because of concerns about utilization rates.

Aim The primary aim of this observational study is to investigate the mid-term effect (1 year) of sit/stand workstations on occupational sitting and standing time as well as the prevalence and intensity of neck and back pain. Secondary aims are the short- and mid-term effects of sit/stand workstations on weekly physical activity as well as daily and weekly sitting and standing time. Furthermore, their effect on the prevalence and intensity of shoulder pain should be analysed. Lastly, predictors for postural changes at work (between sitting and standing) as well as correlates between the IPAQ and OSPAQ questionnaire for office workers should be determinated.

Intervention All employees of an Austrian bank headquarter will be newly equipped with sit/stand workstations by their own company. Prior to this furniture change, all employees were equipped with traditional sit workstations. The study uses the company induced furniture change for scientific purposes. Hence, the furniture change was not driven by the research institution (university).

Methods Within this study 4 assessment days will be executed. They will be carried out 2 weeks before (baseline) and 3, 6 and 12 months after the furniture change. On each assessment day an online survey will be applied. This survey consists of the International Physical Activity Questionnaire (IPAQ), the Occupational Sitting and Physical Activity Questionnaire (OSPAQ), the Nordic Musculoskeletal Questionnaire (NMQ), Visual Analogue Scale (VAS) and well as questions addressing participants´ characteristics.

ELIGIBILITY:
Inclusion Criteria:

* All office workers from a bank headquarter who are affected by the office furniture change (replacement of traditional sitting work desks by sit/stand workstations)
* People with sufficient German language skills (able to understand the questions of the questionnaires)
* People who gave their written consent to participate prior to involvement in the study

Exclusion Criteria:

* People without an employment at the examined bank headquarter
* People who are not able to use sit/stand workstations due to physical impairments
* People on educational or maternity leave

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People of all genders, between 18 and 65 years of age, working in an Austrian bank headquarter, who are affected by their company´s plans to replace all office workstation desks (non-adjustable) by electric height-adjustable sit/stand workstations with desk-height memory function in March 2019.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in occupational sitting time | baseline, 12 months
  Subjects will report the amount of occupational sitting time by means of the OSPAQ.
  The amount of working hours in the last 7 days will be multiplied by the percentage of time spent sitting at work in the last 7 days to get the overall amount of minutes sitting at work per week.
Changes in occupational standing time | baseline, 12 months
  Subjects will report the amount of occupational standing time by means of the OSPAQ.
  The amount of working hours in the last 7 days will be multiplied by the percentage of time spent standing at work in the last 7 days to get the overall amount of minutes standing at work per week.
Changes in the one year prevalence of neck pain | baseline, 12 months
  Subjects will report the one year prevalence of neck pain by means of the Nordic Musculoskeletal Questionnaire.
Changes in the one year prevalence of back pain | baseline, 12 months
  Subjects will report the one year prevalence of back pain by means of the Nordic Musculoskeletal Questionnaire.
Changes in the average one year neck pain intensity (VAS) | baseline, 12 months
  Subjects will report the one year neck pain intensity by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (no pain) to 100 (heavy pain) points.
Changes in the average one year back pain intensity (VAS) | baseline, 12 months
  Subjects will report the one year neck pain intensity by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (no pain) to 100 (heavy pain) points.

SECONDARY OUTCOMES:
Changes in occupational sitting time | baseline, 3 months, 6 months
  Subjects will report the amount of occupational sitting time by means of the OSPAQ.
  The amount of working hours in the last 7 days will be multiplied by the percentage of time spent sitting at work in the last 7 days to get the overall amount of minutes sitting at work per week.
Changes in occupational standing time | baseline, 3 months, 6 months
  Subjects will report the amount of occupational standing time by means of the OSPAQ.
  The amount of working hours in the last 7 days will be multiplied by the percentage of time spent standing at work in the last 7 days to get the overall amount of minutes standing at work per week.
Changes in the average one year prevalence of shoulder pain | baseline, 12 months
  Subjects will report the one year prevalence of shoulder pain by means of the Nordic Musculoskeletal Questionnaire.
Changes in the average one year shoulder pain intensity (VAS) | baseline, 12 months
  Subjects will report the one year neck pain intensity by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (no pain) to 100 (heavy pain) points.
Changes in the average one week prevalence of neck pain | baseline, 3 months, 6 months, 12 months
  Subjects will report the one week prevalence of neck pain by means of the Nordic Musculoskeletal Questionnaire.
Changes in the average one week prevalence of back pain | baseline, 3 months, 6 months, 12 months
  Subjects will report the one week prevalence of back pain by means of the Nordic Musculoskeletal Questionnaire.
Changes in the average one week prevalence of shoulder pain | baseline, 3 months, 6 months, 12 months
  Subjects will report the one week prevalence of shoulder pain by means of the Nordic Musculoskeletal Questionnaire.
Changes in the average one week neck pain intensity (VAS) | baseline, 3 months, 6 months, 12 months
  Subjects will report the one year neck pain intensity by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (no pain) to 100 (heavy pain) points.
Changes in the average one week back pain intensity (VAS) | baseline, 3 months, 6 months, 12 months
  Subjects will report the one year neck pain intensity by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (no pain) to 100 (heavy pain) points.
Changes in the average one week shoulder pain intensity (VAS) | baseline, 3 months, 6 months, 12 months
  Subjects will report the one year neck pain intensity by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (no pain) to 100 (heavy pain) points.
Changes in daily sitting time | baseline, 3 months, 6 months, 12 months
  Subjects will directly report their daily sitting time in hours per day by means of the IPAQ.
Changes in weekly physical activity | baseline, 3 months, 6 months, 12 months
  Subjects will report their weekly physical activity by means of the IPAQ. The amount of walking, moderate and high intensity physical activities as total time in minutes per day, their metabolic equivalents of task (MET) and the frequency in days per week will be multiplied to assess the overall weekly physical activity in MET minutes per week.
  Physical activities will only be considered if they lasted at least for 10 or more minutes over the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schwartz, MSc BSc, Principal Investigator — University of Applied Sciences for Health Professions Upper Austria
Locations (1):
- University of Applied Sciences for Health Professions Upper Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loyen A, van der Ploeg HP, Bauman A, Brug J, Lakerveld J. European Sitting Championship: Prevalence and Correlates of Self-Reported Sitting Time in the 28 European Union Member States. PLoS One. 2016 Mar 2;11(3):e0149320. doi: 10.1371/journal.pone.0149320. eCollection 2016. PMID 26934701
- [Background] Alkhajah TA, Reeves MM, Eakin EG, Winkler EA, Owen N, Healy GN. Sit-stand workstations: a pilot intervention to reduce office sitting time. Am J Prev Med. 2012 Sep;43(3):298-303. doi: 10.1016/j.amepre.2012.05.027. PMID 22898123
- [Background] Chau JY, Daley M, Dunn S, Srinivasan A, Do A, Bauman AE, van der Ploeg HP. The effectiveness of sit-stand workstations for changing office workers' sitting time: results from the Stand@Work randomized controlled trial pilot. Int J Behav Nutr Phys Act. 2014 Oct 8;11:127. doi: 10.1186/s12966-014-0127-7. PMID 25291960
- [Background] Straker L, Abbott RA, Heiden M, Mathiassen SE, Toomingas A. Sit-stand desks in call centres: associations of use and ergonomics awareness with sedentary behavior. Appl Ergon. 2013 Jul;44(4):517-22. doi: 10.1016/j.apergo.2012.11.001. Epub 2012 Dec 4. PMID 23218118
- [Background] Straker L, Mathiassen SE. Increased physical work loads in modern work--a necessity for better health and performance? Ergonomics. 2009 Oct;52(10):1215-25. doi: 10.1080/00140130903039101. PMID 19787501
- [Background] Hill JO, Wyatt HR, Reed GW, Peters JC. Obesity and the environment: where do we go from here? Science. 2003 Feb 7;299(5608):853-5. doi: 10.1126/science.1079857. PMID 12574618
- [Background] Brown WJ, Miller YD, Miller R. Sitting time and work patterns as indicators of overweight and obesity in Australian adults. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1340-6. doi: 10.1038/sj.ijo.0802426. PMID 14574344
- [Background] Peeters GM, Burton NW, Brown WJ. Associations between sitting time and a range of symptoms in mid-age women. Prev Med. 2013 Feb;56(2):135-41. doi: 10.1016/j.ypmed.2012.12.008. Epub 2012 Dec 19. PMID 23262361
- [Background] van der Ploeg HP, Chey T, Korda RJ, Banks E, Bauman A. Sitting time and all-cause mortality risk in 222 497 Australian adults. Arch Intern Med. 2012 Mar 26;172(6):494-500. doi: 10.1001/archinternmed.2011.2174. PMID 22450936
- [Background] van Uffelen JG, van Gellecum YR, Burton NW, Peeters G, Heesch KC, Brown WJ. Sitting-time, physical activity, and depressive symptoms in mid-aged women. Am J Prev Med. 2013 Sep;45(3):276-81. doi: 10.1016/j.amepre.2013.04.009. PMID 23953353
- [Background] van Uffelen JG, Wong J, Chau JY, van der Ploeg HP, Riphagen I, Gilson ND, Burton NW, Healy GN, Thorp AA, Clark BK, Gardiner PA, Dunstan DW, Bauman A, Owen N, Brown WJ. Occupational sitting and health risks: a systematic review. Am J Prev Med. 2010 Oct;39(4):379-88. doi: 10.1016/j.amepre.2010.05.024. PMID 20837291
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Breaks in sedentary time: beneficial associations with metabolic risk. Diabetes Care. 2008 Apr;31(4):661-6. doi: 10.2337/dc07-2046. Epub 2008 Feb 5. PMID 18252901
- [Background] Kerr J, Takemoto M, Bolling K, Atkin A, Carlson J, Rosenberg D, Crist K, Godbole S, Lewars B, Pena C, Merchant G. Two-Arm Randomized Pilot Intervention Trial to Decrease Sitting Time and Increase Sit-To-Stand Transitions in Working and Non-Working Older Adults. PLoS One. 2016 Jan 6;11(1):e0145427. doi: 10.1371/journal.pone.0145427. eCollection 2016. PMID 26735919
- [Background] Peddie MC, Bone JL, Rehrer NJ, Skeaff CM, Gray AR, Perry TL. Breaking prolonged sitting reduces postprandial glycemia in healthy, normal-weight adults: a randomized crossover trial. Am J Clin Nutr. 2013 Aug;98(2):358-66. doi: 10.3945/ajcn.112.051763. Epub 2013 Jun 26. PMID 23803893